CLINICAL TRIAL: NCT02491827
Title: Adjoint Intra-operative Confocal Laser Endomicroscopy (CLE) to Present Tissue on the Cellular Level in Defined Lesions of the Central Nervous System (CNS) During Medically Induced Neurosurgery in Subcranial Tumors and Glioma
Brief Title: Confocal Laser Endomicroscopy (CLE) During Medically Induced Neurosurgery in Craniobasal and Glioma Tumours
Acronym: Cleopatra
Status: Terminated | Type: Observational
Why Stopped: Study stopped by local authorities
Sponsor: Charalampaki, Cleopatra, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: CLE 001
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Tumors
Keywords: optical biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cellvizio mini laser probe: Cellvizio mini laser probe will be administered via the endoscopic device used for the neurosurgical procedure to provide confocal laser endomicroscopy in patients requiring neurosurgery due to glioma multiforme or subcranial tumors
  Interventions: Other: Cellvizio mini laser probe

INTERVENTIONS:
Other: Cellvizio mini laser probe — Cellvizio mini laser probe is administered via the endoscopic device used during the neurosurgical procedures to provide the optical biopsy

SUMMARY:
Purpose of the study is to answer the question whether confocal laser endomicroscopy (CLE, also named 'optical biopsy') might improve the results of medically necessary neurosurgery to prove practicability, safety and harmlessness of CLE during neurosurgical procedures

DETAILED DESCRIPTION:
In patients requiring neurosurgical oncological Intervention using endoscopic devices, a mini laser probe will be administered through the endoscopic device to characterize in vivo the tissue by thousandfold magnification down to the cellular level (so-called optical biopsy). Magnification is presented to the neurosurgeon in time to better differentiate between healthy and pathological tissue. Post-surgery results of in-vivo Differentiation will then be compared to histocytopathological findings.

ELIGIBILITY:
Inclusion Criteria:

* patients administered to the department of neurosurgery requiring neurosurgery due to either diagnosed gliomata (40 patients) or diagnosed subcranial tumors adjacent to or already invading neuronal structures (20 patients)
* patients having given informed consent

Exclusion Criteria:

* severe concomitant diseases probably negatively influencing the participation in this clinical trial
* cardial infarction or stroke within the preceding 12 months
* Treatment resistant hypertonus (systolic blood pressure >200 mmHg or diastolic blood pressure >120 mmHg or a combination of both
* Pulmonic diseases that might result in an advanced risk for anesthetic measurements
* Patients being vaccinated with live vaccines (14 days Prior) or contra Influenza (7 days Prior) to start of the study
* All concomitant findings that might increase in the eyes of the investigator the risk of participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from either subcranial Tumors or cerebral gliomata
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
post-surgery comparison of in-vivo tissue characterization with ex-vivo histocytopathology | duration of hospital stay, an expected average of 7 days

SECONDARY OUTCOMES:
proof of complete removal of pathologic tissue within healthy tissue | during surgical procedure, an expected average time of three hours
optimal tumour remission or reduction after 3 months post-surgery proven by respective diagnostic measurements | 3 months post surgery
Composite measure of missing iatrogenic damage of healthy neuronal structures and preservation of functionality of healthy tissue | individual post-surgery controls, an expected average of up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Cleopatra Charalampaki, MD Prof, Principal Investigator — Department Neurosurgery, Hospital Koeln-Merheim
Locations (1):
- Clinic of Neurosurgery, Hospital of Cologne, Cologne-Merheim, North Rhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No